CLINICAL TRIAL: NCT02446691
Title: A Phase IV, Open-Label, Multi-Center Study to Evaluate the Safety and the 1-year Persistence of Antibody Response Among Children Who Received 4 Doses of the GSK MenACWY Conjugate Vaccine at 2, 4, 6 and 12 Months of Age in South Korea
Brief Title: Evaluation of Antibody Persistence Following 4 MenACWY Vaccinations
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 205336; V59_75 (Other: Novartis); 2014-005392-90 (EudraCT Number)
Record Dates: First submitted 2015-05-13; First posted 2015-05-18 (Estimated); Results first posted 2019-04-01 (Actual); Last update posted 2019-06-27 (Actual); Status verified 2019-06

CONDITIONS: Infections, Meningococcal
MeSH Terms: conditions — Meningococcal Infections | interventions — MenACWY

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MenACWY Group (Experimental): Healthy male and female infants approximately 2 months (55-89 days) of age on the day of consent, who will receive 4 doses of the GSK MenACWY Conjugate Vaccine, administered intramuscularly at 2,4,6 ad 12 months of age.
  Interventions: Biological: MenACWY

INTERVENTIONS:
Biological: MenACWY — Four Intramuscular doses of MenACWY vaccine at 2, 4, 6 and 12 months of age followed by two blood samples at 13 and 24 months of age.

SUMMARY:
This is Phase IV, Open label, Multicenter study. Subject's parents and/or legal guardian will be provided information about the trial. If interested and if eligible, they will then be asked to provide signed informed consent. The initial study visit can occur immediately after signed informed consent has been obtained. Approximately 135 subjects will be enrolled to receive 4 doses of intramuscular MenACWY vaccine at 2, 4, 6 and 12 months of age.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female 2 month-old infants (55 - 89 days) on the day of consent.
2. Infants whose parents or legal guardians have voluntary given written informed consent after the nature of the study has been explained according to local regulatory requirements, prior to study entry.
3. Infants whose parents or legal guardians can comply with study procedures including follow-up

Exclusion Criteria:

1. Previously received any meningococcal A, C, W and Y vaccines.
2. Previous confirmed or suspected disease caused by N. meningitidis or who have had household contact with and/or intimate exposure to an individual with laboratory confirmed N. meningitidis infection at any time since birth.
3. Progressive, unstable or uncontrolled clinical conditions.
4. A history of anaphylactic shock, asthma, urticaria or other allergic reaction after previous vaccinations or known hypersensitivity to any vaccine component, such as latex allergy.
5. Experienced significant acute or chronic infection within the previous 7 days or have experienced fever (temperature ≥ 38.0°C [100.4°F]) within the previous 3 days.
6. Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
7. Received treatment with systemic administration corticosteroids (PO/IV/IM) for more than 14 consecutive days from birth
8. Ever received blood, blood products and/or plasma derivatives or any parenteral immunoglobulin preparation (including Hepatitis B immune globulin) at any time since birth and for the full length of the study.
9. Any bleeding disorder which is considered as a contraindication to intramuscular injection or blood draw.
10. Any condition which, in the opinion of the investigator, might interfere with the results of the study or pose additional risk to the subject due to participation in the study.
11. Received or are planning to receive any investigational or non-registered medicinal product from birth and throughout the study.
12. Received oral or parenteral antibiotic treatment in the 3 days prior to the scheduled blood draw (topical antibiotics are acceptable, including antibiotic eye drops).
13. Relatives of site research staff working on this study.

Ages: 2 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 128 (Actual)
Dates: Start 2015-07-13 (Actual); Primary Completion 2017-12-28 (Actual); Study Completion 2017-12-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (5):
- South Korea (5):
  - GSK Investigational Site, Ansan-si
  - GSK Investigational Site, Incheon
  - GSK Investigational Site, Jeonju
  - GSK Investigational Site, Seongnam-si
  - GSK Investigational Site, Seoul

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled from 6 centers in South Korea.
Pre-assignment Details: All enrolled subjects were vaccinated.
Groups:
- MenACWY Group: Healthy male and female infants approximately 2 months (55-89 days) of age on the day of consent, who received 4 doses of the GSK MenACWY Conjugate Vaccine, administered intramuscularly, at 2, 4, 6 and 12 months of age.
Period: Overall Study
Arm/Group | MenACWY Group
Started | 128
Completed | 117
Not Completed | 11
Not completed — Withdrawal by Subject | 2
Not completed — Lost to Follow-up | 8
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | MenACWY Group
Number analyzed (Participants) | 128
Age, Continuous [Mean (Standard Deviation); unit: Days] | 71.7 (8.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59
  Male | 69
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 127
  Unspecified | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Any Solicited Adverse Events (AEs) Within 30 Minutes After Each Vaccination.
Description: Solicited signs and symptoms occurring within 30 minutes following each vaccination, include solicited local events (e.g. injection site erythema, induration and tenderness -threshold for Erythema and Induration: Type II- None [<10mm], Any[>=10 mm]), solicited systemic events (e.g. change in eating habits, sleepiness, irritability, vomiting, diarrhea, fever[ body temperature >=38°C measured preferably via tympanic route]), and any other solicited event like use of analgesic/antipyretics for treatment or for prophylaxis
Time Frame: Within 30 minutes of each vaccination
Population: Analysis was performed on the solicited safety set, which included all subjects who received a study vaccination and reported any solicited adverse event data and/or indicators of solicited adverse events.
Measure: Count of Participants; unit: Participants
Arm/Group | MenACWY Group
Number analyzed (Participants) | 128
Participants
  Injection site erythema, Vaccination 1, Any | 0
  Injection site erythema, Vaccination 2, Any | 0
  Injection site erythema, Vaccination 3, Any | 0
  Injection site erythema, Vaccination 4, Any: number analyzed (Participants) | 124
  Injection site erythema, Vaccination 4, Any | 1
  Injection site induration, Vaccination 1, Any | 0
  Injection site induration, Vaccination 2, Any | 0
  Injection site induration, Vaccination 3, Any | 0
  Injection site induration, Vaccination 4, Any: number analyzed (Participants) | 124
  Injection site induration, Vaccination 4, Any | 1
  Injection site tenderness, Vaccination 1, Any | 0
  Injection site tenderness, Vaccination 2, Any | 0
  Injection site tenderness, Vaccination 3, Any | 0
  Injection site tenderness, Vaccination 4, Any: number analyzed (Participants) | 124
  Injection site tenderness, Vaccination 4, Any | 0
  Change in eating habits, Vaccination 1, Any | 0
  Change in eating habits, Vaccination 2, Any | 0
  Change in eating habits, Vaccination 3, Any | 0
  Change in eating habits, Vaccination 4, Any: number analyzed (Participants) | 124
  Change in eating habits, Vaccination 4, Any | 0
  Diarrhea, Vaccination 1, Any | 0
  Diarrhea, Vaccination 2, Any | 0
  Diarrhea, Vaccination 3, Any | 0
  Diarrhea, Vaccination 4, Any: number analyzed (Participants) | 124
  Diarrhea, Vaccination 4, Any | 0
  Irritability, Vaccination 1, Any | 0
  Irritability, Vaccination 2, Any | 0
  Irritability, Vaccination 3, Any | 0
  Irritability, Vaccination 4, Any: number analyzed (Participants) | 124
  Irritability, Vaccination 4, Any | 0
  Sleepiness, Vaccination 1, Any | 0
  Sleepiness, Vaccination 2, Any | 0
  Sleepiness, Vaccination 3, Any | 0
  Sleepiness, Vaccination 4, Any: number analyzed (Participants) | 124
  Sleepiness, Vaccination 4, Any | 0
  Vomiting, Vaccination 1, Any | 0
  Vomiting, Vaccination 2, Any | 0
  Vomiting, Vaccination 3, Any | 0
  Vomiting, Vaccination 4, Any: number analyzed (Participants) | 124
  Vomiting, Vaccination 4, Any | 1
  Fever, Vaccination 1, Yes | 0
  Fever, Vaccination 1, No | 128
  Fever, Vaccination 2, Yes | 0
  Fever, Vaccination 2, No | 128
  Fever, Vaccination 3, Yes | 0
  Fever, Vaccination 3, No | 128
  Fever, Vaccination 4, Yes: number analyzed (Participants) | 124
  Fever, Vaccination 4, Yes | 0
  Fever, Vaccination 4, No: number analyzed (Participants) | 124
  Fever, Vaccination 4, No | 124

2. Primary Outcome: Number of Subjects With Any Solicited Local AEs From Day 1 to Day 7 After Each Vaccination
Description: Solicited local AEs reported from day 1 to day 7 after each vaccination were assessed. Assessed local symptoms include injection site erythema, injection site induration and injection site tenderness. Any = incidence of a particular symptom regardless of intensity grade.Threshold for Erythema and Induration: Type II None (<10 mm), Any (>=10 mm)
Time Frame: From Day 1 to Day 7 after each vaccination
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | MenACWY Group
Number analyzed (Participants) | 128
Participants
  Injection site erythema, Vaccination 1, Any | 4
  Injection site erythema, Vaccination 2, Any | 6
  Injection site erythema, Vaccination 3, Any: number analyzed (Participants) | 127
  Injection site erythema, Vaccination 3, Any | 6
  Injection site erythema, Vaccination 4, Any: number analyzed (Participants) | 124
  Injection site erythema, Vaccination 4, Any | 6
  Injection site induration, Vaccination 1, Any | 4
  Injection site induration, Vaccination 2, Any | 9
  Injection site induration, Vaccination 3, Any: number analyzed (Participants) | 127
  Injection site induration, Vaccination 3, Any | 3
  Injection site induration, Vaccination 4, Any: number analyzed (Participants) | 124
  Injection site induration, Vaccination 4, Any | 6
  Injection site tenderness, Vaccination 1, Any | 17
  Injection site tenderness, Vaccination 2, Any | 21
  Injection site tenderness, Vaccination 3, Any: number analyzed (Participants) | 127
  Injection site tenderness, Vaccination 3, Any | 14
  Injection site tenderness, Vaccination 4, Any: number analyzed (Participants) | 124
  Injection site tenderness, Vaccination 4, Any | 20

3. Primary Outcome: Number of Subjects With Any Solicited Systemic AEs From Day 1 to Day 7 After Each Vaccination.
Description: Solicited systemic AEs reported from day 1 to day 7 after each vaccination were assessed. Assessed systemic symptoms include change in eating habits, sleepiness, irritability, vomiting, diarrhea and fever (body temperature ≥ 38°C (100.4°F)).
Time Frame: From Day 1 to Day 7 after each vaccination
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | MenACWY Group
Number analyzed (Participants) | 128
Participants
  Change in eating habits, Vaccination 1, Any | 29
  Change in eating habits, Vaccination 2, Any | 21
  Change in eating habits, Vaccination 3, Any: number analyzed (Participants) | 127
  Change in eating habits, Vaccination 3, Any | 21
  Change in eating habits, Vaccination 4, Any: number analyzed (Participants) | 124
  Change in eating habits, Vaccination 4, Any | 24
  Diarrhea, Vaccination 1, Any | 15
  Diarrhea, Vaccination 2, Any | 13
  Diarrhea, Vaccination 3, Any: number analyzed (Participants) | 127
  Diarrhea, Vaccination 3, Any | 15
  Diarrhea, Vaccination 4, Any: number analyzed (Participants) | 124
  Diarrhea, Vaccination 4, Any | 17
  Irritability, Vaccination 1, Any | 58
  Irritability, Vaccination 2, Any | 49
  Irritability, Vaccination 3, Any: number analyzed (Participants) | 127
  Irritability, Vaccination 3, Any | 47
  Irritability, Vaccination 4, Any: number analyzed (Participants) | 124
  Irritability, Vaccination 4, Any | 45
  Sleepiness, Vaccination 1, Any | 52
  Sleepiness, Vaccination 2, Any | 31
  Sleepiness, Vaccination 3, Any: number analyzed (Participants) | 127
  Sleepiness, Vaccination 3, Any | 28
  Sleepiness, Vaccination 4, Any: number analyzed (Participants) | 124
  Sleepiness, Vaccination 4, Any | 20
  Vomiting, Vaccination 1, Any | 26
  Vomiting, Vaccination 2, Any | 20
  Vomiting, Vaccination 3, Any: number analyzed (Participants) | 127
  Vomiting, Vaccination 3, Any | 15
  Vomiting, Vaccination 4, Any: number analyzed (Participants) | 124
  Vomiting, Vaccination 4, Any | 5
  Fever, Vaccination 1, Yes | 4
  Fever, Vaccination 1, No | 124
  Fever, Vaccination 2, Yes | 10
  Fever, Vaccination 2, No | 118
  Fever, Vaccination 3, Yes: number analyzed (Participants) | 127
  Fever, Vaccination 3, Yes | 6
  Fever, Vaccination 3, No: number analyzed (Participants) | 127
  Fever, Vaccination 3, No | 121
  Fever, Vaccination 4, Yes: number analyzed (Participants) | 124
  Fever, Vaccination 4, Yes | 15
  Fever, Vaccination 4, No: number analyzed (Participants) | 124
  Fever, Vaccination 4, No | 109

4. Primary Outcome: Number of Subjects With Any Medically Attended Unsolicited AEs and AEs Leading to Premature Withdrawal
Description: An unsolicited adverse event is an adverse event that was not solicited using a Subject Diary and that was spontaneously communicated by a subject parent(s)/legal guardian(s)] who has signed the informed consent. All medically attended unsolicited AEs were collected from Day 1 to Visit 6.
Time Frame: From Day 1 to Visit 6 (at 24 Months of age)
Population: Analysis was performed on the unsolicited safety set, which included all subjects who received a study vaccination and reported any unsolicited adverse event data.
Measure: Count of Participants; unit: Participants
Arm/Group | MenACWY Group
Number analyzed (Participants) | 128
Participants
  Any Medically Attended Unsolicited AEs | 85
  AEs leading to premature withdrawal | 0

5. Primary Outcome: Number of Subjects With Serious AEs (SAEs)
Description: Subjects reporting SAEs from day 1 to visit 6 (at 24 months of age) were assessed. A serious adverse event (SAE) is defined as any untoward medical occurrence that at any dose results in one or more of the following: death, is life-threatening, required or prolonged hospitalization, persistent or significant disability/incapacity, congenital anomaly/or birth defect, An important and significant medical event that may not be immediately life threatening or resulting in death or hospitalization but, based upon appropriate medical judgment, may jeopardize the subject or may require intervention to prevent one of the other outcomes listed above.
Time Frame: From Day 1 to Visit 6 (At 24 months of age)
Population: Analysis was performed on the overall safety set, which included all subjects who received a study vaccination and reported any solicited/unsolicited adverse event data.
Measure: Count of Participants; unit: Participants
Arm/Group | MenACWY Group
Number analyzed (Participants) | 128
Participants | 26

6. Primary Outcome: Percentage of Subjects With Human Serum Bactericidal Assay (hSBA) Titers ≥ 8 Against Each N.Meningitidis Serogroup A,C,W and Y at 24 Months of Age.
Description: To assess antibody persistence against N. meningitidis serogroups A, C, W and Y at 1 year after completion of a 4-dose infant vaccination series (2, 4, 6 and 12 months of age) of MenACWY vaccine as measured by serum bactericidal assay using human serum complement.
Time Frame: At 24 months of age (Visit 6)
Population: Analysis was performed on the Full analysis set (FAS), which included all enrolled subjects who received at least one study vaccination and provided an evaluable hSBA Visit 6 assessment, one year after completion of a 4-dose infant vaccination series (2, 4, 6 and 12 months of age), for at least one serogroup.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | MenACWY Group
Number analyzed (Participants) | 114
Percentage of subjects
  Serogroup A | 39 [30.4 to 49.1]
  Serogroup C: number analyzed (Participants) | 110
  Serogroup C | 61 [51.1 to 70.1]
  Serogroup W: number analyzed (Participants) | 113
  Serogroup W | 88 [80.1 to 93.1]
  Serogroup Y | 89 [81.3 to 93.8]

7. Primary Outcome: Percentage of Subjects With Rabbit Serum Bactericidal Assay (rSBA) Titers ≥ 8, Against Each N.Meningitidis Serogroup at 24 Months of Age
Description: To assess antibody persistence against N. Meningitidis serogroups A, C, W and Y at 1 year after completion of a 4-dose infant vaccination series (2, 4, 6 and 12 months of age) of MenACWY vaccine as measured by serum bactericidal assay using rabbit serum complement
Time Frame: At 24 months of age (Visit 6)
Population: Analysis was performed on the FAS, which included all enrolled subjects who receive at least one study vaccination and provided an evaluable rSBA Visit 6 assessment, one year after completion of a 4-dose infant vaccination series (2, 4, 6 and 12 months of age), for at least one serogroup.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | MenACWY Group
Number analyzed (Participants) | 108
Percentage of subjects
  Serogroup A | 99 [94.9 to 99.98]
  Serogroup C | 54 [43.8 to 63.3]
  Serogroup W | 69 [59.8 to 77.9]
  Serogroup Y: number analyzed (Participants) | 107
  Serogroup Y | 90 [82.3 to 94.8]

8. Primary Outcome: Percentage of Subjects With Rabbit Serum Bactericidal Assay (rSBA) Titers ≥ 128 Against Each N.Meningitidis Serogroup at 24 Months of Age
Description: as for outcome 7
Time Frame: At 24 months of age (Visit 6)
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | MenACWY Group
Number analyzed (Participants) | 108
Percentage of subjects
  Serogroup A | 98 [93.5 to 99.77]
  Serogroup C | 30 [21.2 to 39.2]
  Serogroup W | 62 [52.2 to 71.2]
  Serogroup Y: number analyzed (Participants) | 107
  Serogroup Y | 80 [71.6 to 87.4]

9. Secondary Outcome: Percentage of Subjects With hSBA ≥8 Against Each N. Meningitidis Serogroups A, C, W and Y at 13 Months of Age
Description: To assess antibody response against N. meningitidis serogroups A, C, W and Y at 1 month after completion of a 4-dose infant vaccination series (2, 4, 6 and 12 months of age) of MenACWY vaccine as measured by serum bactericidal assay using human serum complement.
Time Frame: At 13 months of age (Visit 5)
Population: The Analysis was done on FAS hSBA 1 month, which included all enrolled subjects who received at least one study vaccination and who provided evaluable hSBA immunogenicity data at 1 month after last vaccination for at least one serogroup.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | MenACWY Group
Number analyzed (Participants) | 122
Percentage of subjects
  Serogroup A | 94 [88.5 to 97.7]
  Serogroup C | 98 [94.2 to 99.80]
  Serogroup W | 100 [97.0 to 100.0]
  Serogroup Y: number analyzed (Participants) | 120
  Serogroup Y | 100 [97.0 to 100.0]

10. Secondary Outcome: Percentage of Subjects With rSBA Titers ≥ 8 Against Each N. Meningitidis Serogroups A, C, W and Y at 13 Months of Age
Description: To assess antibody response against N. meningitidis serogroups A, C, W and Y at 1 month after completion of a 4-dose infant vaccination series (2, 4, 6 and 12 months of age) of MenACWY vaccine as measured by serum bactericidal assay using rabbit serum complement.
Time Frame: At 13 months of age (Visit 5)
Population: The Analysis was done on FAS rSBA 1 month, which included all enrolled subjects who received atleast one study vaccination and who provided evaluable rSBA immunogenicity data at 1 month after last vaccination for atleast one serogroup.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | MenACWY Group
Number analyzed (Participants) | 116
Percentage of subjects
  Serogroup A: number analyzed (Participants) | 115
  Serogroup A | 100 [96.8 to 100.0]
  Serogroup C: number analyzed (Participants) | 115
  Serogroup C | 99 [95.3 to 99.98]
  Serogroup W: number analyzed (Participants) | 115
  Serogroup W | 100 [96.8 to 100.0]
  Serogroup Y | 100 [96.9 to 100.0]

11. Secondary Outcome: Percentage of Subjects With rSBA Titers ≥ 128 Against Each N. Meningitidis Serogroups A, C, W and Y at 13 Months of Age
Description: as for outcome 10
Time Frame: At 13 months of age (Visit 5)
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | MenACWY Group
Number analyzed (Participants) | 116
Percentage of subjects
  Serogroup A: number analyzed (Participants) | 115
  Serogroup A | 100 [96.8 to 100.0]
  Serogroup C: number analyzed (Participants) | 115
  Serogroup C | 92 [85.7 to 96.4]
  Serogroup W: number analyzed (Participants) | 115
  Serogroup W | 98 [93.9 to 99.79]
  Serogroup Y | 98 [93.9 to 99.79]

12. Secondary Outcome: hSBA Geometric Mean Titers (GMTs) Against Each N. Meningitidis Serogroups A, C, W and Y at 24 Months of Age
Description: To assess persistence of antibody response in terms of GMTs using hSBA assay against N. meningitidis serogroups A, C, W and Y at 1 year after completion of a 4-dose infant vaccination series (2, 4, 6 and 12 months of age) of MenACWY vaccine.
Time Frame: At 24 months of age (Visit 6)
Population: Analysis was performed on the Full analysis set (FAS), which included all enrolled subjects who received atleast one study vaccination and provided an evaluable hSBA Visit 6 assessment, one year after completion of a 4-dose infant vaccination series (2, 4, 6 and 12 months of age ), for atleast one serogroup.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | MenACWY Group
Number analyzed (Participants) | 114
Titers
  Serogroup A | 6.80 [5.19 to 8.93]
  Serogroup C: number analyzed (Participants) | 110
  Serogroup C | 13.04 [9.65 to 17.63]
  Serogroup W: number analyzed (Participants) | 113
  Serogroup W | 53.56 [40.42 to 70.97]
  Serogroup Y | 50.75 [38.76 to 66.45]

13. Secondary Outcome: rSBA GMTs Against Each N. Meningitidis Serogroups A, C, W and Y at 24 Months of Age
Description: To assess persistence of antibody response in terms of GMTs using rSBA assay against N. meningitidis serogroups A, C, W and Y at 1 year after completion of a 4-dose infant vaccination series (2, 4, 6 and 12 months of age) of MenACWY vaccine.
Time Frame: At 24 months of age (Visit 6)
Population: Analysis was performed on the Full analysis set (FAS), which included all enrolled subjects who received atleast one study vaccination and provided an evaluable rSBA Visit 6 assessment, one year after completion of a 4-dose infant vaccination series (2, 4, 6 and 12 months of age ), for atleast one serogroup.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | MenACWY Group
Number analyzed (Participants) | 108
Titers
  Serogroup A | 2269.48 [1761.12 to 2924.59]
  Serogroup C | 17.17 [11.28 to 26.14]
  Serogroup W | 114.04 [65.22 to 199.39]
  Serogroup Y: number analyzed (Participants) | 107
  Serogroup Y | 310.91 [203.23 to 475.65]

14. Secondary Outcome: hSBA GMTs Against Each N. Meningitidis Serogroups A, C, W and Y at 13 Months of Age
Description: To assess antibody response in terms of GMTs using hSBA assay against N. meningitidis serogroups A, C, W and Y at 1 month after completion of a 4-dose infant vaccination series (2, 4, 6 and 12 months of age) of MenACWY vaccine.
Time Frame: At 13 months of age (Visit 5)
Population: The Analysis was done on FAS hSBA 1 month, which included all enrolled subjects who received atleast one study vaccination and provided evaluable hSBA immunogenicity data at 1 month after last vaccination for atleast one serogroup.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | MenACWY Group
Number analyzed (Participants) | 122
Titers
  Serogroup A | 107.90 [85.73 to 135.81]
  Serogroup C | 201.04 [157.90 to 255.96]
  Serogroup W | 426.74 [338.34 to 538.24]
  Serogroup Y: number analyzed (Participants) | 120
  Serogroup Y | 359.39 [280.59 to 460.31]

15. Secondary Outcome: rSBA GMTs Against Each N. Meningitidis Serogroups A, C, W and Y at 13 Months of Age.
Description: To assess antibody response in terms of GMTs using rSBA assay against N. meningitidis serogroups A, C, W and Y at 1 month after completion of a 4-dose infant vaccination series (2, 4, 6 and 12 months of age) of MenACWY vaccine.
Time Frame: At 13 months of age (Visit 5)
Population: The Analysis was done on FAS rSBA 1 month, which included all enrolled subjects who received atleast one study vaccination and provided evaluable rSBA immunogenicity data at 1 month after last vaccination for atleast one serogroup.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | MenACWY Group
Number analyzed (Participants) | 116
Titers
  Serogroup A: number analyzed (Participants) | 115
  Serogroup A | 7394.18 [6057.42 to 9025.93]
  Serogroup C: number analyzed (Participants) | 115
  Serogroup C | 735.07 [545.22 to 991.03]
  Serogroup W: number analyzed (Participants) | 115
  Serogroup W | 2718.69 [2031.77 to 3637.85]
  Serogroup Y | 2226.70 [1731.21 to 2863.99]

ADVERSE EVENTS:
Time Frame: Solicited local and systemic adverse events (AEs): from Day 1 to Day 7 after each vaccination. Unsolicited AEs, serious AEs (SAEs): From Day 1 to study end (visit 6).
Arm/Group | MenACWY Group
All-Cause Mortality (participants affected / at risk) | 0/128
Serious Adverse Events (participants affected / at risk) | 26/128
Other Adverse Events (participants affected / at risk) | 112/128
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MenACWY Group (N=128)
Buried penis syndrome (Congenital, familial and genetic disorders) | 1 (1)
Enteritis (Gastrointestinal disorders) | 1 (1)
Bronchiolitis (Infections and infestations) | 5 (6)
Croup infectious (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Hand-foot-and-mouth disease (Infections and infestations) | 1 (1)
Herpangina (Infections and infestations) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1)
Pharyngotonsillitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 4 (5)
Pneumonia influenzal (Infections and infestations) | 1 (1)
Pneumonia parainfluenzae viral (Infections and infestations) | 1 (1)
Pneumonia respiratory syncytial viral (Infections and infestations) | 1 (1)
Pneumonia viral (Infections and infestations) | 1 (1)
Tonsillitis (Infections and infestations) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 3 (3)
Viral infection (Infections and infestations) | 1 (1)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1)
Tendon injury (Injury, poisoning and procedural complications) | 1 (1)
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MenACWY Group (N=128)
Hydrocele (Congenital, familial and genetic disorders) | 1 (1)
Tympanic membrane perforation (Ear and labyrinth disorders) | 1 (1)
Eye discharge (Eye disorders) | 2 (2)
Retinal disorder (Eye disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 41 (178)
Enteritis (Gastrointestinal disorders) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 2 (2)
Mouth ulceration (Gastrointestinal disorders) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (2)
Vomiting (Gastrointestinal disorders) | 42 (168)
Atopy (Immune system disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1)
Adenovirus infection (Infections and infestations) | 1 (1)
Bronchiolitis (Infections and infestations) | 11 (14)
Bronchitis (Infections and infestations) | 11 (21)
Cellulitis (Infections and infestations) | 1 (1)
Croup infectious (Infections and infestations) | 3 (3)
Ear infection (Infections and infestations) | 1 (1)
Enterovirus infection (Infections and infestations) | 3 (4)
Exanthema subitum (Infections and infestations) | 3 (3)
Gastroenteritis (Infections and infestations) | 9 (10)
Gastroenteritis viral (Infections and infestations) | 1 (1)
Gianotti-Crosti syndrome (Infections and infestations) | 1 (1)
Hand-foot-and-mouth disease (Infections and infestations) | 6 (6)
Herpangina (Infections and infestations) | 1 (1)
Hordeolum (Infections and infestations) | 1 (1)
Impetigo (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 15 (18)
Oral candidiasis (Infections and infestations) | 1 (1)
Otitis externa (Infections and infestations) | 1 (1)
Otitis media (Infections and infestations) | 5 (5)
Otitis media acute (Infections and infestations) | 11 (13)
Parainfluenzae virus infection (Infections and infestations) | 1 (1)
Pharyngitis (Infections and infestations) | 3 (3)
Pharyngotonsillitis (Infections and infestations) | 6 (6)
Pneumonia (Infections and infestations) | 5 (7)
Respiratory tract infection viral (Infections and infestations) | 1 (1)
Rhinitis (Infections and infestations) | 6 (7)
Sinusitis (Infections and infestations) | 2 (3)
Tonsillitis (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 32 (52)
Viral infection (Infections and infestations) | 4 (4)
Concussion (Injury, poisoning and procedural complications) | 4 (4)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Ear canal injury (Injury, poisoning and procedural complications) | 1 (1)
Eye contusion (Injury, poisoning and procedural complications) | 1 (1)
Foreign body in gastrointestinal tract (Injury, poisoning and procedural complications) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1)
Lip injury (Injury, poisoning and procedural complications) | 2 (2)
Radial head dislocation (Injury, poisoning and procedural complications) | 1 (2)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1)
Skull fracture (Injury, poisoning and procedural complications) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (7)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 (9)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 3 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 4 (4)
Pityriasis alba (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 3 (3)
Urticaria (Skin and subcutaneous tissue disorders) | 3 (4)
Injection site pain (General disorders) | 41 (136)
Pyrexia (General disorders) | 33 (68)
Injection site induration (General disorders) | 22 (67)
Injection site erythema (General disorders) | 16 (40)
Hypophagia (Metabolism and nutrition disorders) | 59 (230)
Somnolence (Nervous system disorders) | 67 (265)
Irritability (Psychiatric disorders) | 86 (461)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2015-08-25): https://cdn.clinicaltrials.gov/large-docs/91/NCT02446691/Prot_000.pdf
  • Statistical Analysis Plan (2016-06-07): https://cdn.clinicaltrials.gov/large-docs/91/NCT02446691/SAP_001.pdf